CLINICAL TRIAL: NCT03292640
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group, Vehicle-Controlled Study of the Safety and Efficacy of DFD-03 Lotion in the Treatment of Acne Vulgaris for 12 Weeks
Brief Title: A Study of the Safety and Efficacy of DFD-03 Lotion in the Treatment of Acne Vulgaris for 12 Weeks
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DFD-03-CD-006
Record Dates: First submitted 2017-09-21; First posted 2017-09-25 (Actual); Results first posted 2020-06-09 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — tazarotene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DFD-03 Lotion (0.1% tazarotene) (Experimental): DFD-03 Lotion (0.1% tazarotene)
  Interventions: Drug: DFD-03 (0.1% tazarotene) Lotion
- DFD-03 Vehicle (0% tazarotene) (Placebo Comparator): DFD-03 Vehicle Lotion (0% tazarotene)
  Interventions: Drug: DFD-03 (0% tazarotene) Lotion (Placebo)

INTERVENTIONS:
Drug: DFD-03 (0.1% tazarotene) Lotion — DFD-03 Lotion (0.1% tazarotene) - twice daily application
  Other Names: DFD-03
  Arms: DFD-03 Lotion (0.1% tazarotene)
Drug: DFD-03 (0% tazarotene) Lotion (Placebo) — DFD-03 Vehicle Lotion (0% tazarotene) - twice daily application
  Other Names: Placebo
  Arms: DFD-03 Vehicle (0% tazarotene)

SUMMARY:
Enrollment of subjects with mild to moderate facial acne vulgaris.

Co-Primary efficacy endpoints included:

* Absolute change from Baseline to Week 12 in the inflammatory lesion counts on the face
* Absolute change from Baseline to Week 12 in the non-inflammatory lesion counts on the face
* Proportion of subjects with a clinical response of "success" at Week 12 for lesions on the face. Success based on IGA is defined as an IGA score of 0 (Clear) or 1 (Almost clear) at Week 12 with at least a 2-grade reduction from Baseline.

DETAILED DESCRIPTION:
Enrollment of subjects with mild to moderate facial acne vulgaris. Acne lesions of any severity on the chest and/or back (including shoulders) were enrolled provided they had mild to moderate acne on the face. During the 12-week treatment period subjects used the study product twice daily with approximately 12 hours between applications. Subjects were instructed to treat the entire face (and chest/back including shoulders, if applicable).

Co-Primary efficacy endpoints included:

* Absolute change from Baseline to Week 12 in the inflammatory lesion counts on the face
* Absolute change from Baseline to Week 12 in the non-inflammatory lesion counts on the face
* Proportion of subjects with a clinical response of "success" at Week 12 for lesions on the face. Success based on IGA is defined as an IGA score of 0 (Clear) or 1 (Almost clear) at Week 12 with at least a 2-grade reduction from Baseline.

The primary safety endpoint was treatment-emergent adverse events (TEAEs). Other safety variables included local cutaneous tolerance evaluation (dryness, non-lesional erythema, peeling, stinging, burning, and itching) and vital signs (blood pressure and pulse rate). Urine pregnancy tests were performed at Baseline and at every visit through Week 12 for all female subjects. A physical examination was performed at the Baseline Visit.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 9 years of age.
2. Female subjects must be having their period at the Baseline Visit (as reported by the subject), except for subjects using hormonal contraceptives that preclude menstrual periods, if the subject is premenarcheal, is postmenopausal for at least 12 months prior to baseline, is surgically sterilized (i.e. tubal ligation) or if the subject is without a uterus and /or both ovaries.
3. A clinical diagnosis of facial mild to moderate acne vulgaris. Subjects with acne lesions on the chest and/or back (including shoulders) in addition to those on the face have the option of treating their back and/or chest (including shoulders) in addition to their face.
4. Inflammatory lesion count (papules and pustules) of at least 20 on the face, and non-inflammatory lesion count (closed and open comedones) of at least 25 on the face, including the nose, and no more than 2 nodulocystic lesions on the face, including the nose.
5. Females, regardless of childbearing potential:

   Must have a negative urine pregnancy test and if sexually active, must be on or use an acceptable method of birth control.
6. Subjects must be willing to comply with sun avoidance measures for the face (as well as back/chest and shoulders, if applicable) including use of investigator-approved sunscreen and/or hats, have limited sun exposure time, and have no tanning bed use.
7. Subject must be in good general health as determined by the investigator and supported by the medical history, physical examination, and normal or not clinically significant abnormal vital signs (blood pressure and pulse).

Exclusion Criteria:

1. Females who are pregnant or lactating or planning to become pregnant during the study period.
2. Treatment with the following products:

   1. Topical acne treatments or other topical facial medication on the treatment area in the 14 days prior to the Baseline Visit, including prescription and non-prescription products.
   2. Systemic corticosteroids, systemic acne treatments including systemic antibiotics used for treatment of acne, potential photosensitizing agents spironolactone, flutamide, or immunosuppressant drugs in the 30 days prior to the Baseline Visit.
   3. Systemic retinoid use in the 180 days prior to the Baseline Visit.
   4. Undertaken certain facial procedures such as chemical peel, laser treatment, photodynamic therapy, acne surgery, cryodestruction or chemodestruction, x-ray therapy, intralesional steroids, dermabrasion, or depilation (except eyebrow shaping) in the 30 days prior to the Baseline Visit. After the subject is enrolled in the study, eyebrow shaping (except for tweezing) is prohibited.
   5. Treatment with a medication or procedure that, in the opinion of the investigator, would put the subject at unacceptable risk for participation in the study or may interfere with evaluations in the study.
   6. Treatment with an investigational product or device in the 30 days prior to the Baseline Visit.
3. Known allergic reaction to retinoids or tazarotene or any of the other ingredients of these products.
4. Presence of any facial skin disease or condition that would interfere with the study or place the subject at unacceptable risk including sunburn, rosacea, seborrheic dermatitis, perioral dermatitis, lupus, dermatomyositis, psoriasis, eczema, squamous cell carcinoma, acneiform eruptions caused by medications, steroid acne, steroid folliculitis, bacterial folliculitis or any other facial disease or condition.
5. Subjects with a serious and/or chronic medical condition such as chronic or active liver disease, renal impairment, heart disease, severe respiratory disease, rheumatoid arthritis, current malignancies, immunocompromised conditions, or any other disease that, in the opinion of the investigator, would interfere with the study or place the subject at unacceptable risk.

7. Subjects who have been treated for alcohol dependence or alcohol or drug abuse in the year.

8. Subjects who have been in another investigational trial within 30 days.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 547 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2018-05-14 (Actual); Study Completion 2018-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas R. Sidgiddi, M.D., Study Director — Dr. Reddy's Laboratories
Locations (1):
- Center for Dermatology Clinical Research Inc., Fremont, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- DFD-03 Lotion (0.1% Tazarotene): DFD-03 (0.1% tazarotene) Lotion: Subjects will apply a quarter (U.S coin) size amount of the study product all over the moistened face and rub it into the skin until foamy. Care should be taken to avoid the areas around the eyes, mouth, and nostrils. After a short time, the subject will rinse off the product by thoroughly rinsing with warm water. This procedure will be followed twice daily, in the morning and at bedtime, approximately 12 hours apart.
- DFD-03 Vehicle (0% Tazarotene): DFD-03 (0% tazarotene) Lotion (Placebo): Subjects will apply a quarter (U.S coin) size amount of the study product all over the moistened face and rub it into the skin until foamy. Care should be taken to avoid the areas around the eyes, mouth, and nostrils. After a short time, the subject will rinse off the product by thoroughly rinsing with warm water. This procedure will be followed twice daily, in the morning and at bedtime, approximately 12 hours apart.
Period: Overall Study
Arm/Group | DFD-03 Lotion (0.1% Tazarotene) | DFD-03 Vehicle (0% Tazarotene)
Started | 275 | 272
Completed | 214 | 230
Not Completed | 61 | 42
Not completed — Withdrawal by Subject | 17 | 16
Not completed — Adverse Event | 20 | 2
Not completed — Lost to Follow-up | 24 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DFD-03 Lotion (0.1% Tazarotene) | DFD-03 Vehicle (0% Tazarotene) | Total
Number analyzed (Participants) | 275 | 272 | 547
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 93 | 85 | 178
  Between 18 and 65 years | 182 | 187 | 369
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.7 (6.5) | 21.3 (7.6) | 21.0 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 143 | 111 | 254
  Male | 132 | 161 | 293
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 28 | 32 | 60
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  Black or African American | 45 | 40 | 85
  White | 186 | 186 | 372
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 12 | 24
Region of Enrollment [Number; unit: participants]
  United States | 275 | 272 | 547

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in the Inflammatory Lesion Counts on the Face
Description: Change in inflammatory lesion counts on the face from baseline to Week 12
Time Frame: Baseline to Week 12
Population: Intent To Treat (ITT) Population - All subjects randomized and dispensed study medication.
Measure: Mean (Standard Deviation); unit: Lesions
Units Other Than Participants: Face
Arm/Group | DFD-03 Lotion (0.1% Tazarotene) | DFD-03 Vehicle (0% Tazarotene)
Number analyzed (Participants) | 275 | 272
Number analyzed (Face) | 275 | 272
Lesions
  Baseline | 29.4 (13.82) | 29.7 (13.27)
  Week 12 | 15.9 (12.14) | 18.2 (16.58)

2. Primary Outcome: Proportion of Subjects With a Clinical Response of "Success" at Week 12 for Lesions on the Face Based on IGA.
Description: IGA success at Week 12 (an IGA score of 0 (Clear) or 1 (almost clear) with at least a 2-grade reduction from baseline)
Time Frame: Baseline to Week 12
Population: Intent To Treat (ITT) Population - All subjects randomized and dispensed study medication.
Measure: Count of Participants; unit: Participants
Groups:
- DFD-03 Lotion (0.1% Tazarotene): DFD-03 (0.1% tazarotene) Lotion: Subjects applied a quarter (U.S coin) size amount of the study product all over the moistened face and rub it into the skin until foamy. After a short time, the subject rinsed off the product with warm water. This procedure was followed twice daily, in the morning and at bedtime, approximately 12 hours apart.
- DFD-03 Vehicle (0% Tazarotene): DFD-03 (0% tazarotene) Lotion (Placebo): Subjects applied a quarter (U.S coin) size amount of the study product all over the moistened face and rub it into the skin until foamy. After a short time, the subject rinsed off the product with warm water. This procedure was followed twice daily, in the morning and at bedtime, approximately 12 hours apart.
Arm/Group | DFD-03 Lotion (0.1% Tazarotene) | DFD-03 Vehicle (0% Tazarotene)
Number analyzed (Participants) | 275 | 272
Participants | 58 | 26

3. Primary Outcome: Absolute Change in the Non-inflammatory Lesion Counts on the Face
Description: Change in non-inflammatory lesion counts on the face from baseline to Week 12 - will be analyzed using the ANCOVA model
Time Frame: Baseline to Week 12
Population: Intent To Treat (ITT) Population - All subjects randomized and dispensed study medication
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | DFD-03 Lotion (0.1% Tazarotene) | DFD-03 Vehicle (0% Tazarotene)
Number analyzed (Participants) | 275 | 272
Lesions
  Baseline | 44.8 (33.93) | 44.4 (27.75)
  Week 12 | 24.3 (18.13) | 29.7 (23.12)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time treatment was initiated until study product treatment was discontinued (i.e. up to 12 weeks), except for spontaneously reported SAEs, which were to be reported up to 30 days after discontinuing study product use.
Groups:
- DFD-03 Lotion (0.1% Tazarotene): DFD-03 (0.1% tazarotene) Lotion was to be applied twice daily for 12 weeks
- DFD-03 Vehicle (0% Tazarotene): DFD-03 Vehicle Lotion (0% tazarotene) was to be applied twice daily for 12 weeks
Arm/Group | DFD-03 Lotion (0.1% Tazarotene) | DFD-03 Vehicle (0% Tazarotene)
All-Cause Mortality (participants affected / at risk) | 0/275 | 0/272
Serious Adverse Events (participants affected / at risk) | 2/275 | 0/272
Other Adverse Events (participants affected / at risk) | 0/275 | 0/272
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFD-03 Lotion (0.1% Tazarotene) (N=275) | DFD-03 Vehicle (0% Tazarotene) (N=272)
Auto Accident with head trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stomach Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-02): https://cdn.clinicaltrials.gov/large-docs/40/NCT03292640/Prot_SAP_000.pdf